CLINICAL TRIAL: NCT04223258
Title: Automatic Oxygen Control for Reducing Extremes of Oxygen Saturation (AreOS): A Randomised Control Trial
Acronym: AreOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Collaborators: Vyaire Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 277057
Record Dates: First submitted 2020-01-03; First posted 2020-01-10 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Prematurity
Keywords: Preterm Infants; Automatic oxygen control; Respiratory support
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Oxygen Control (Experimental): Infants randomized to this arm will be monitored using automatic oxygen control system on the ventilator. When infants oxygen saturation are out of the target range the ventilator will adjust the oxygen delivery depending on the saturation of the infant to bring the saturation int he target range.
  Interventions: Device: Automatic Oxygen control
- Manual oxygen control (Active Comparator): Infants randomized to this arm will be receive oxygen delivery adjustments manually by the nursing and medical team taking care of the infants. When the infants oxygen saturation are out of the target range, the staff will manually adjust the oxygen delivery.
  Interventions: Other: Manual Oxygen Control

INTERVENTIONS:
Device: Automatic Oxygen control — The CLiO device is integral to the Avea infant ventilator and allows automated OXYGEN adjustment aiming to maintain SpO2 within assigned target range using neonatal pulse oximeter. When first started it adopts the FiO2 previously set by the clinician as the initial 'Baseline FiO2' level. Thereafter, the changes to the FiO2 and their frequency depend on whether SpO2 is below, above or within the target range, the trend in SpO2 and all changes are proportionate to the 'Baseline FiO2' level.
  Arms: Automatic Oxygen Control
Other: Manual Oxygen Control — In the manual arm the oxygen is adjusted manually by the clinical team.
  Arms: Manual oxygen control

SUMMARY:
Oxygen treatment is common in babies born early (preterm) and requiring intensive care. Having too much or too little oxygen can increase the risk of damage to the eyes and lungs, and contribute to death or disability. Preterm infants because of their immaturity experience episodes of low oxygen levels. The low oxygen episodes are primarily due to pauses in their breathing (Apnoea of prematurity) and immaturity of their lung. These episodes persist for weeks. The lower the gestation at birth the longer the duration of these events. Studies have shown that these episodes of low oxygen saturations especially if frequent and prolonged is associated with poor developmental outcome, severe eye disease and lung disease.

Traditionally, the oxygen delivery is manually adjusted when infant has low oxygen saturation. However previous studies have shown despite the best efforts the oxygen level can only be maintained less than half of the time and nearly a one-fifth of the time infant spends in low oxygen levels and nearly one third of the time in high oxygen levels. Now it is possible to maintain oxygen level in target range by using automatic control of oxygen delivery. With the proposed study, we would like to study the efficacy of automatic control of oxygen delivery in reducing the time spent in low oxygen levels.

DETAILED DESCRIPTION:
Supplemental oxygen remains by far the most commonly used 'drug' in neonatal intensive care units. The goal of oxygen therapy is to maintain normal oxygenation while minimizing hypoxemia and hypoxemia. Preterm infants are particularly vulnerable to oxygen toxicity and oxidative stress leading to retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), and periventricular leukomalacia (PVL)[1]. It's also well known that preterm infants experience hypoxic events which are primarily linked to cardiovascular instability and apnea of prematurity. These events vary as the infant matures. Martin R et al showed in their study that these hypoxic events peaked around 2-4 weeks and decreases by 6-8 weeks in preterm infants (2). Exposure to prolonged and frequent hypoxemic episodes has been associated with increased morbidity and mortality [3-5]. Prolonged hypoxic events (Saturation less than 80% for more than 1 minute) have been associated with severe ROP and impaired neurodevelopmental outcome in survivors (2, 5).

Peripheral oxygen saturation monitoring is standard of care in preterm infants. Traditionally oxygen saturation (SpO2) targeting is carried out by manual adjustment of fraction of inspired oxygen (FiO2) by the caregiver based on the monitored oxygen saturation. However, in practice this is only partially achieved during routine care[6]. Hagadorn et al conducted a study in 14 centers and showed that preterm infants under 28 weeks' gestation receiving oxygen spent on average only 48% of the time with SpO2 within the prescribed target range, about 36% of the time above and 16% of the time with SpO2 below the target range [7].

Preterm infants have frequent fluctuations in SpO2 due to their cardio-respiratory instability requiring frequent adjustments of FiO2 [7]. Consequently, these particularly vulnerable infants spend significant time with SpO2 outside intended range and are often exposed to extremes of hypoxemia and hyperoxaemia. It is now possible to have automated control of inspired oxygen using a device (CLiO2™) incorporated in Avea® ventilator. The device continuously monitors the oxygen saturation and adjusts the oxygen delivery to maintain oxygen saturation within the target range. The safety, feasibility and efficacy of this device have already been established [9-14]. There has been further improvement in the algorithm of the pulse oximeter incorporated in Avea® ventilator to achieve a better normative distribution around the median SpO2 value[15]. Automated control of FiO2 significantly improves compliance of oxygen saturation targeting and significantly reduces exposure to hypoxemia as well as hyperoxaemia [9-14, 16,]. Automatic control of oxygen delivery is available in both invasive and non-invasive mode of ventilation (17). The Avea ventilators are equipped with Automatic Oxygen control with invasive as well as non-invasive mode of ventilation.

Previous studies looking at the efficacy of automated oxygen control mostly have been a crossover model and the study duration less than 48 hours. As previously mentioned, preterm infants experience hypoxic events for few weeks before cardiopulmonary maturation is established. Hence, it's important to study these events over a longer period of time. The objective of this randomised controlled trial is to evaluate the efficacy of the automatic oxygen control function in reducing the time spent in extremes of oxygen saturations (less than 80%), in preterm infants for the entire period of their respiratory support on invasive or non-invasive mode of ventilation.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants less than 33 weeks (23+0 to 32+6 weeks)

• Receiving invasive or non-invasive mode of respiratory support

Exclusion Criteria:

* Infants more than or equal to 33 weeks
* Preterm infants with congenital anomalies
* Infants on a non-conventional mode of invasive or non-invasive ventilation

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
proportion of time spent in extreme saturation ( less than or equal to 80%) | Through study completion, an average of 8 weeks
  The primary outcome of this study is proportion of time spent in extreme saturation (less than or equal to 80%) in preterm infants <33 weeks receiving invasive or non-invasive form of respiratory support.

SECONDARY OUTCOMES:
Proportion of time spent in target saturation | Through study completion, an average of 8 weeks
  Proportion of the time spent in target saturation of 90-95%
Proportion of time spent in saturation more than or equal to 98% | Through study completion, an average of 8 weeks
  The proportion of time spent in more than or equal to 98% through the entire period of respiratory support
Number of episodes of prolonged hypoxemia (SpO2 less than 80% for more than 60 sec) | Through study completion, an average of 8 weeks
  Toatal number of episodes of prolonged hypoxemia through the respiratory support
Brochopulmonary Dysplasia at 36 weeks PMA | Upto 36 weeks post menstrual age
  Oxygen supplementation or need for respiratory support at 36 weeks PMA
Oxygen need at day 28 | 4 weeks
  Need for oxygen on day 28
Severe Retinopathy of Prematurity | Upto 36 weeks post menstrual age
  Severe ROP requiring treatment
Periventricular Leuckomalacia | Upto 36 weeks post menstrual age
  PVL diagnosed by Brain imaging through their stay in the NICU
Total number of days on supplemental oxygen less than 30% | Upto 36 weeks post menstrual age
  The total number of days the infant has spent in the oxygen less than 30%
Length of hospital day | Upto 36 weeks post menstrual age
  Total duration of stay in Neonatal Unit

CONTACTS AND LOCATIONS:
Overall Officials: Vrinda Nair, MD,FRCPCH, Principal Investigator — South Tees NHS trust
Locations (1):
- South Tees NHS Trust, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Martin RJ, Wang K, Koroglu O, Di Fiore J, Kc P. Intermittent hypoxic episodes in preterm infants: do they matter? Neonatology. 2011;100(3):303-10. doi: 10.1159/000329922. Epub 2011 Oct 3. PMID 21986336
- [Background] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Carlo WA, Finer NN, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Schibler K, Newman NS, Ambalavanan N, Frantz ID 3rd, Piazza AJ, Sanchez PJ, Morris BH, Laroia N, Phelps DL, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Ehrenkranz RA, Watterberg KL, Higgins RD. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1959-69. doi: 10.1056/NEJMoa0911781. Epub 2010 May 16. PMID 20472937
- [Background] Stenson B, Brocklehurst P, Tarnow-Mordi W; U.K. BOOST II trial; Australian BOOST II trial; New Zealand BOOST II trial. Increased 36-week survival with high oxygen saturation target in extremely preterm infants. N Engl J Med. 2011 Apr 28;364(17):1680-2. doi: 10.1056/NEJMc1101319. No abstract available. PMID 21524227
- [Background] Poets CF, Roberts RS, Schmidt B, Whyte RK, Asztalos EV, Bader D, Bairam A, Moddemann D, Peliowski A, Rabi Y, Solimano A, Nelson H; Canadian Oxygen Trial Investigators. Association Between Intermittent Hypoxemia or Bradycardia and Late Death or Disability in Extremely Preterm Infants. JAMA. 2015 Aug 11;314(6):595-603. doi: 10.1001/jama.2015.8841. PMID 26262797
- [Background] Laptook AR, Salhab W, Allen J, Saha S, Walsh M. Pulse oximetry in very low birth weight infants: can oxygen saturation be maintained in the desired range? J Perinatol. 2006 Jun;26(6):337-41. doi: 10.1038/sj.jp.7211500. PMID 16598294
- [Background] Hagadorn JI, Furey AM, Nghiem TH, Schmid CH, Phelps DL, Pillers DA, Cole CH; AVIOx Study Group. Achieved versus intended pulse oximeter saturation in infants born less than 28 weeks' gestation: the AVIOx study. Pediatrics. 2006 Oct;118(4):1574-82. doi: 10.1542/peds.2005-0413. PMID 17015549
- [Derived] Nair V, Kannan Loganathan P, Lal MK, Pringleton H, Bachman TE, Brodlie M, Dixon P. Automatic oxygen control for reducing extremes of oxygen saturation: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2023 Mar;108(2):136-141. doi: 10.1136/archdischild-2022-324160. Epub 2022 Aug 23. PMID 35999043